CLINICAL TRIAL: NCT02802007
Title: Pilot Trial of the Elipse™ Intragastric Balloon System for the Treatment of Overweight and Obese Individuals
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Allurion Technologies (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TRL-1000-0001-B
Record Dates: First submitted 2016-04-12; First posted 2016-06-16 (Estimated); Last update posted 2016-06-16 (Estimated); Status verified 2016-06

CONDITIONS: Obesity; Overweight
MeSH Terms: conditions — Obesity; Overweight

ARMS (1):
- Elipse Intragastric Balloon (Experimental): Patients seeking weight loss received the Elipse Intragastric Balloon.
  Interventions: Device: Elipse Intragastric Balloon

INTERVENTIONS:
Device: Elipse Intragastric Balloon

SUMMARY:
This is a prospective, non-randomized, open trial to be conducted in overweight and obese individuals. The primary objective is to evaluate the safety of the Elipse™ Intragastric Balloon System for the treatment of overweight and obese individuals. The secondary objective is to collect efficacy and device performance information to assist with future trial design and device iterations.

ELIGIBILITY:
Inclusion Criteria:

* Patient, female or male, 18 to 64 years of age.
* Patient must be able to understand and be willing to sign an IC document.
* Patient must be willing to participate in all aspects of the trial for the duration of the trial.
* Patient must be motivated to lose weight and have realistic expectations.
* Patient must complete the screening requirement to complete one week of Daily Eating Diaries and Daily Weight Logs.
* Patient must pass the Screening Behavioral Interview.
* Patient must understand that even though they undergo the Elipse™ Treatment, they must follow the physician guidelines for eating behaviors and lifestyle modifications for weight loss.
* Patient has a BMI of ≥ 27.0.
* Females must be willing to use contraception throughout the course of the trial until they exit.
* Patients must have a primary care physician that follows them for any co-morbid conditions.
* Patients must live within 160 kilometers of the trial site and not plan to move out of the vicinity for the trial duration.
* Patients must be fully ambulatory without any chronic orthopedic disease or reliance on crutches, walkers or a wheelchair that could preclude exercise during the trial.
* Patient must have a stable home environment that is supportive of the patient's efforts to lose weight.
* If Patient is an ex-smoker, they must be an ex-smoker for more than a year.
* Patient agrees to refrain from any reconstructive and/or cosmetic surgery that may affect body weight during the study such as mammoplasty and lipoplasty.

Exclusion Criteria:

* Patient has symptomatic congestive heart failure, cardiac arrhythmia or unstable coronary artery disease.
* Patient has pre-existing respiratory disease such as chronic obstructive pulmonary disease (COPD), pneumonia or cancer.
* Female subject who is pregnant (i.e., has a positive urine or blood pregnancy test prior to surgery), is suspected to be pregnant, is lactating or is of childbearing potential but refuses to use adequate contraception during the study.
* Patient has had previous bariatric or gastric surgery.
* Patient has a history of acute pancreatitis.
* Patient has a history of small bowel obstructions.
* Patients with a history of abdominal and/or pelvic surgery EXCLUDING only ONE of the following surgeries that was performed at least 12 months prior to the Elipse™ Treatment: cesarean section, diagnostic laparoscopy, laparoscopic appendectomy, laparoscopic cholecystectomy. (For example: if a patient has had 2 cesarean sections, or one cesarean section and a laparoscopic appendectomy they would be excluded. If a patient had one cesarean section they may be included.)
* Patient has history of/or signs and/or symptoms of esophageal, gastric, or duodenal disease including but not limited to hiatal hernias >2 centimeter (cm), inflammatory diseases, cancer, and varices.
* Patient has a specific diagnosed genetic or hormonal cause for obesity such as hypothyroidism or PraderWilli syndrome.
* Patient has poorly controlled diabetes.
* Patient has renal and/or hepatic insufficiency.
* Patient has systemic infection or abscess at the site to be treated.
* Patient is undergoing chronic steroid therapy.
* Patient is undergoing immunosuppressive therapy.
* Patient is presently taking heparin, coumadin, warfarin, or other anticoagulants or other medications which impede coagulation or platelet aggregation.
* Patient is unable or unwilling to discontinue use of aspirin and/or non-steroidal anti-inflammatory agents (NSAIDs) at least 14 days prior to treatment and continuing for 14 days post-treatment.
* Patient has a history of pulmonary embolism or blood coagulation disorders.
* Patient is unable to discontinue either prescription or over the counter weight loss medications at least 30 days prior to treatment and continuing for the remainder of the trial
* Patient has cardiac pacemaker or other electric implantable device.
* Patient has a history of using any tobacco products including but not limited to cigars, cigarettes, and pipes within 12 months prior to enrollment.
* Patient has poorly controlled psychiatric disease such as depression.
* Patient has eating disorders including night eating syndrome (NES), Bulimia, or binge eating disorder, or who continuously graze on food for the majority of the day.
* Patient has uncontrolled life stressors at baseline such as divorce, or illness/death of personal acquaintances.
* Patient currently uses or has a history of illicit drug use or excessive alcohol use.
* Patient has participated in a clinical study with an investigational new drug, biological, or therapeutic device within ≤ 28 days prior to enrollment in this trial, and does not agree to abstain from participation in other clinical trials of any kind during this trial.
* Patient is not of sufficient medical health as determined by the PI to participate in the trial.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2014-08; Primary Completion 2016-07 (Estimated)

PRIMARY OUTCOMES:
The occurrence and frequency of adverse events (AE)s, adverse device effects (ADE)s, serious adverse events (SAE)s, serious adverse device effects (SADE)s and unanticipated serious adverse device effects (USADE)s. | 4 months

SECONDARY OUTCOMES:
Change in weight: Percent Excess Weight Loss (%EWL) | 4 months
Change in weight: Total Body Weight Loss (kg) | 4 months
Change in weight: Percent Total Body Weight Loss (%TBWL) | 4 months

CONTACTS AND LOCATIONS:
Locations (2):
- Ostrava University Hospital, Ostrava, Czechia
- Iatriko Palaiou Faliro, Athens, Greece